CLINICAL TRIAL: NCT03272165
Title: A Randomized, Double-blind, Placebo-controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single Ascending Doses of MEDI1341 in Healthy Male and Female Volunteers
Brief Title: Single Ascending Dose Study of MEDI1341 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Covance (Industry); MMS Holdings, Inc (Unknown); Catalent (Industry); Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6340C00001
Record Dates: First submitted 2017-06-29; First posted 2017-09-05 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Parkinson's Disease
Keywords: Healthy Volunteers; Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Immunogenicity
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants are randomized to one of two groups within a cohort of 8 participants (N=6 MEDI1341; N=2 placebo)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Placebo (Placebo Comparator): Participants will receive a single intravenous (IV) infusion of placebo matched to MEDI1341 and will be followed up for 13 weeks.
  Interventions: Drug: Placebo
- Cohort 1: MEDI1341 Dose 1 (Experimental): Participants will receive a single IV infusion of MEDI1341 Dose 1 and will be followed up for 13 weeks.
  Interventions: Drug: MEDI1341
- Cohort 2: MEDI1341 Dose 2 (Experimental): Participants will receive a single IV infusion of MEDI1341 Dose 2 and will be followed up for 13 weeks.
  Interventions: Drug: MEDI1341
- Cohort 3: MEDI1341 Dose 3 (Experimental): Participants will receive a single IV infusion of MEDI1341 Dose 3 and will be followed up for 13 weeks.
  Interventions: Drug: MEDI1341
- Cohort 4: MEDI1341 Dose 4 (Experimental): Participants will receive a single IV infusion of MEDI1341 Dose 4 and will be followed up for 13 weeks.
  Interventions: Drug: MEDI1341
- Cohort 5: MEDI1341 Dose 5 (Experimental): Participants will receive a single IV infusion of MEDI1341 Dose 5 and will be followed up for 13 weeks.
  Interventions: Drug: MEDI1341
- Cohort 6: MEDI1341 Dose 6 (Experimental): Participants will receive a single IV infusion of MEDI1341 Dose 6 and will be followed up for 13 weeks.
  Interventions: Drug: MEDI1341

INTERVENTIONS:
Drug: MEDI1341 — Participants will receive IV infusion of MEDI1341 doses as stated in the arms' description.
  Other Names: TAK-341
  Arms: Cohort 1: MEDI1341 Dose 1; Cohort 2: MEDI1341 Dose 2; Cohort 3: MEDI1341 Dose 3; Cohort 4: MEDI1341 Dose 4; Cohort 5: MEDI1341 Dose 5; Cohort 6: MEDI1341 Dose 6
Drug: Placebo — Participants will receive IV infusion of placebo matched to MEDI1341.
  Arms: Placebo

SUMMARY:
This is a study of single ascending intravenous doses of MEDI1341 or placebo in up to 48 healthy volunteers, aged 18 to 65 years. The study will include up to 6 planned cohorts; each cohort will comprise 8 participants.

Each participant will receive a single 60 minute intravenous infusion of MEDI1341 or placebo and will undergo scheduled assessments over a period of 13 weeks.

The main aim of the study is to assess the safety and tolerability of single doses of MEDI1341 in healthy volunteers.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled study of single ascending intravenous doses of MEDI1341 in male and nonfertile female healthy volunteers, aged 18 to 65 years.

The study will include up to 6 planned cohorts; each cohort will comprise 8 participants. Within each cohort, 6 participants will be randomized to receive MEDI1341 and 2 will be randomized to receive placebo. A Safety Review Committee will review data from each cohort before progression to the next higher dose cohort occurs. On Day 1, each randomized participant will receive a single 60 minute intravenous infusion of MEDI1341 or placebo and will undergo scheduled safety, pharmacokinetic, pharmacodynamic, and immunogenicity assessments. Additional study assessments will occur on Days 2, 4, 8, 15, 22, 29, 43, 57, and 92.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy, with no clinically significant abnormality identified on the medical or laboratory evaluation at screening
* Participants must weigh ≥50 kg and must have a body mass index between 18 and 32 kg/m^2, inclusive
* Participants must have a 12-lead electrocardiogram recorded at screening that is normal for the appropriate age group and shows no abnormalities that will compromise safety in this study
* Participants must have no clinically significant findings on the clinical neurological examinations at screening and at baseline or on the ophthalmic examination at screening.

Exclusion Criteria:

* Nicotine use within 6 months before screening
* Considered to be at a high risk of developing a stroke
* Significant medical history of dizziness, blackouts, fainting, or vaso-vagal attacks
* History of any significant ophthalmic disorder, including congenital, genetic or acquired conditions affecting the retina or choroid
* History of severe allergy or history of hypersensitivity to immunizations or immunoglobulins
* History of any significant psychiatric disorder
* History of alcohol abuse
* History of cancer within 5 years of screening
* History of drug abuse
* Any contraindication to Lumbar Puncture
* Any clinically significant abnormality in ECG rhythm, conduction or morphology
* Positive serologic findings at screening for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen, or hepatitis C virus antibodies
* Use of prescription or non-prescription drugs
* For female participants, a positive serum or urine pregnancy test result at screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs) | Day 1 through 92 days after a single dose of study drug
  An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Number of Participants With Abnormal Vital Signs, Physical and Neurological Examinations, and Body Weight Measurements Reported as TEAEs | Day 1 through 92 days after a single dose of study drug
  Vital signs assessment included body temperature, respiration rate, pulse rate, and blood pressure. Participants with abnormal vital signs, physical and neurological examinations, and body weight measurements reported as TEAEs are reported.
Change from Baseline in 12-Lead Electrocardiogram (ECG) Data in Paper and Digital Recordings (PR Interval, QRS Duration, QT Interval, QTcF Interval, and RR Interval) | 12-lead paper ECG: Baseline (Day -49) to Day 92; Digital ECG: Baseline (Day 1) to Day 92
  Changes from baseline in 12-Lead ECG data in paper recordings (PR interval, QRS duration, QT interval, and QTcF interval) and digital recordings (PR interval, QRS duration, QT interval, QTcF interval, and RR interval) are reported.
Change from Baseline in Heart Rate by 12-Lead ECG in Paper and Digital Recordings | 12-lead paper ECG: Baseline (Day -49) to Day 92; Digital ECG: Baseline (Day 1) to Day 92
  Change from baseline in heart rate by 12-Lead ECG in paper and digital recordings are reported.
Number of Participants With Abnormal Laboratory Parameters Reported as TEAEs | Day 1 through 92 days after a single dose of study drug
  Laboratory assessment included hematology, clinical chemistry, and urinalysis. Participants with abnormal laboratory parameters reported as TEAEs are reported.
Number of Abnormal Findings for Ophthalmic Assessment (Ophthalmic Examination and Slit-lamp Examination) for Placebo and Cohorts 4 to 6 at Follow-up Visit | Follow-up Visit (Day 57)
  Number of abnormal findings for ophthalmic assessment (ophthalmic examination and slit-lamp examination) at follow-up visit (Day 57) are reported.
Intraocular Pressure at Screening for Placebo and Cohorts 4 to 6 | Screening (Day -49)
  Intraocular pressure at Screening (Day -49) is reported.
Intraocular Pressure at Day 29 for Placebo and Cohorts 4 to 6 | Day 29
  Intraocular pressure at Day 29 is reported.
Intraocular Pressure at Day 92 for Placebo and Cohorts 4 to 6 | Day 92
  Intraocular pressure at Day 92 is reported.
Number of Participants With Injection Site Reactions | Day 1
  Participants who had injection site reactions (bleeding, bruising, erythema, swelling, or induration) on Day 1 are reported.
Visual Analogue Scale (VAS) Pain Score for Site Reaction Pain | Day 1 (within 24 hours after end of infusion)
  The VAS (0 to 10 cm) was used to describe reaction site pain. The score 0 means 'no pain at all' and 10 score means 'worst pain imaginable'. The higher the VAS score, the greater the reaction site pain experienced.
Number of Participants With Suicidal Ideation and Suicidal Behavior Assessed by Columbia Suicide Severity Rating Scale (C-SSRS) | Screening (Day -49) through 92 days after a single dose of study drug
  The C-SSRS is a scale capturing occurrence, severity, and frequency of suicide-related thoughts and behaviours, and has a binary response (yes/no).
  * Suicidal Ideation: a "yes" answer to any one of 5 suicidal ideation questions: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intent to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent.
  * Suicidal Behaviour: a "yes" answer to any of 5 suicidal behaviour questions: preparatory acts or behaviour, aborted attempt, interrupted attempt, actual attempt (non-fatal), completed suicide.
Number of Participants With Montreal Cognitive Assessment (MoCA) Total Score at Screening (Day -1) | Screening (Day -1)
  The MoCA is s standardized cognitive screening tool for mild cognitive impairment and dementia. The total score was used as outcome measure and this score ranges from 0-31, with higher scores representing better cognitive ability and scores below 26 were considered as cognitive dysfunction.
Number of Participants With MoCA Total Score at Day 92 | Day 92
  The MoCA is s standardized cognitive screening tool for mild cognitive impairment and dementia. The total score was used as outcome measure and this score ranges from 0-31, with higher scores representing better cognitive ability and scores below 26 were considered as cognitive dysfunction.

SECONDARY OUTCOMES:
Maximum Observed Serum Concentration (Cmax) of MEDI1341 | Day 1 (predose; 0 minute and 8 and 24 hours at the end of infusion), and Days 4, 8, 15, 22, 29, 43, 57, and 92
  The Cmax of MEDI1341 is reported.
Time to Maximum Serum Concentration (tmax) of MEDI1341 | Day 1 (predose; 0 minute and 8 and 24 hours at the end of infusion), and Days 4, 8, 15, 22, 29, 43, 57, and 92
  The tmax of MEDI1341 is reported.
Area Under the Serum Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUC0-t) of MEDI1341 | Day 1 (predose; 0 minute and 8 and 24 hours at the end of infusion), and Days 4, 8, 15, 22, 29, 43, 57, and 92
  The AUC0-t of MEDI1341 is reported.
Area Under the Concentration-time Curve From Time 0 to Infinity (AUC0-∞) of MEDI1341 | Day 1 (predose; 0 minute and 8 and 24 hours at the end of infusion), and Days 4, 8, 15, 22, 29, 43, 57, and 92
  The AUC0-∞ of MEDI1341 is reported.
Terminal Half-life (t1/2λz) of MEDI1341 | Day 1 (predose; 0 minute and 8 and 24 hours at the end of infusion), and Days 4, 8, 15, 22, 29, 43, 57, and 92
  The t1/2λz of MEDI1341 is reported.
Serum Clearance (CL) of MEDI1341 | Day 1 (predose; 0 minute and 8 and 24 hours at the end of infusion), and Days 4, 8, 15, 22, 29, 43, 57, and 92
  The CL of MEDI1341 is reported.
Volume of Distribution at Steady State (Vss) of MEDI1341 | Day 1 (predose; 0 minute and 8 and 24 hours at the end of infusion), and Days 4, 8, 15, 22, 29, 43, 57, and 92
  The Vss of MEDI1341 is reported.
Mean Residence Time (MRT) of MEDI1341 | Day 1 (predose; 0 minute and 8 and 24 hours at the end of infusion), and Days 4, 8, 15, 22, 29, 43, 57, and 92
  The MRT of MEDI1341 is reported.
Percentage Change From Baseline in Plasma Concentrations of Total α-synuclein | Baseline (Day 1 predose) through Day 92
  Maximum change from baseline through Day 92 and change from baseline at Day 92 in plasma concentrations of total α-synuclein are reported.
Percentage Change From Baseline in Cerebrospinal Fluid Concentrations of Free α-synuclein | Baseline (Day 1 predose) and Day 29
  Change from baseline in cerebrospinal fluid concentrations of free α-synuclein is reported.
Percentage of Participants With Positive Antidrug Antibodies (ADAs) to MEDI1341 by Titer Levels at Day 92 | Day 92
  Percentage of participants with positive ADAs to MEDI1341 by titer levels are reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanelle Kam, MD, CPI, Principal Investigator — Covance Dallas CRU, USA; John E Blanchard, MD, Principal Investigator — Covance Madison CRU, USA
Locations (2):
- United States (2):
  - Research Site, Dallas, Texas
  - Research Site, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymised individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved, AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsor tool. Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home